CLINICAL TRIAL: NCT01965834
Title: Phase II Study to Evaluate Fenofibrate Therapy in Patients With Smoldering or Symptomatic Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of adequate accrual.
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Denise Pereira, Assistant Professor of Clinical, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20110069
Record Dates: First submitted 2013-10-15; First posted 2013-10-18 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Fenofibrate
MeSH Terms: conditions — Multiple Myeloma | interventions — Fenofibrate; fenofibric acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fenofibrate Therapy (Experimental): Fenofibrate orally daily for each 28 day cycle, per study protocol.
  Interventions: Drug: Fenofibrate

INTERVENTIONS:
Drug: Fenofibrate — Upon screening, registration and enrollment, all subjects will receive Fenofibrate 160 mg orally daily for at least 2 months and may continue receiving study medication for as long as in the opinion of the investigator there is clinical benefit in doing so. Patients with calculated creatinine clearance < 50 mL/min will receive a reduced dose of 54 mg orally daily.
  Other Names: Fenofibric acid

SUMMARY:
Multiple myeloma cells are dependent on calcium (Ca2+) for their function. Specifically, Ca2+ is required for the function of the endoplasmic reticulum in which proteins, including immunoglobulins, are folded prior to their release from the cell. Multiple myeloma cells secrete large concentrations of immunoglobulins continuously and as result depend on mitochondria activity to replenish the Ca2+ levels in the endoplasmic reticulum as was shown in vitro in our lab. Fenofibrate has been shown to inhibit mitochondrial function resulting in inhibition of protein folding in the endoplasmic reticulum of multiple myeloma (MM) cells that leads to the induction of a stress signal known as the unfolded protein response and subsequently apoptosis. The effective anti-myeloma concentrations for fenofibrate are attainable in the clinical setting as they are in the same range as the effective concentrations for anti-hyperlipidemic effect. The investigators propose to evaluate fenofibrate therapy in multiple myeloma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have histologically or cytologically confirmed multiple myeloma (smoldering myeloma and symptomatic multiple myeloma).
2. Patients must have measurable disease and therefore must have at least one of the following:

   * Serum M-protein ≥ 1 gm/dL (≥ 10 gm/L)
   * Urine M-protein ≥ 200 mg/24 hr
   * Serum free light chain (FLC) assay: involved FLC ≥ 10 mg/dL (≥ 100 mg/L) provided serum FLC ratio is abnormal.
3. Male or female ≥ 18 years of age.
4. Life expectancy of ≥ 6 months.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
6. Normal organ and marrow function as defined below:

   * Absolute Neutrophil Count (ANC) ≥ 1,000/mm^3
   * Platelets ≥75,000/mm^3
   * Hemoglobin ≥ 8 g/dL
   * Calculated serum creatinine (calculated by Cockcroft-Gault method) ≥ 30 mL/min
   * Aspartate transaminase (AST)/serum glutamic oxaloacetic transaminase (SGOT)/ Alanine transaminase (ALT)/serum glutamate-pyruvate transaminase (SGPT) ≤ 2.5 X upper limit of normal (ULN)
   * Total bilirubin ≤ 1.5 X ULN
7. Patient must be at least 2 weeks from prior chemotherapy, radiation therapy, biological therapy, immunotherapy, major surgery and any other investigational anti-cancer therapy prior to the first dose of study drug.
8. Patient has recovered from toxicities (≤ Grade 2) and/or complications from prior therapy.
9. Patient is able to swallow capsules and is able to take or tolerate oral medications on a continuous basis.
10. Female patients of childbearing potential must be willing to use 2 adequate barrier methods of contraception to prevent pregnancy or agrees to abstain from heterosexual intercourse for at least 1 month before dosing, and while women are on study and for up to 12 weeks after last dose of study drug. Adequate contraceptive methods include intrauterine device, diaphragm with spermicide, cervical cap with spermicide, or female condom with spermicide. Spermicides alone are not an acceptable method of contraception.
11. Male patients agree to have female partners of childbearing potential use 2 adequate barrier methods of contraception as described in Section 3.1.10.
12. Female patients of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose of study drug.
13. Patient is available for periodic blood sampling, study related assessments and management at the treating institution for the duration of the study.
14. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients who only present with isolated plasmacytomas
2. Inability to swallow oral medication.
3. Prior allogeneic stem cell transplant (subject with prior autologous transplant is eligible).
4. Patient has plans to undergo any type of stem cell transplantation (allogeneic or autologous) within 4 weeks of initiation of study therapy.
5. Concurrent therapy with 3-hydroxy-3-methyl-glutaryl-coenzyme A reductase (HMG-CoA) Reductase Inhibitors.
6. Patient with gallbladder disease or cholelithiasis.
7. Patient has active liver disease, including biliary cirrhosis and unexplained liver function abnormalities.
8. Patients receiving renal dialysis.
9. History of hypersensitivity to fenofibrate or fenofibric acid, including sever skin rashes (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis)
10. Patients who would be receiving any other investigational agents while on study.
11. Participation in any investigational drug study within 4 weeks preceding the start of study treatment.
12. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
13. Patient has systemic infection requiring treatment.
14. Patient has acute diffuse infiltrative pulmonary disease or pericardial disease.
15. Subject is receiving corticosteroid therapy (> 10 mg of prednisone or equivalent).
16. Subject is a regular user or has a recent history (within the last year) of any illicit drugs, or substance abuse.
17. Subject is pregnant or breast feeding, or expecting to conceive or father children within the projected duration of the study.
18. Subject is known to be HIV positive.
19. Subject has clinically active Hepatitis B or C
20. History of prior malignancy except for cervical carcinoma in situ, non-melanoma skin cancer, adequately treated localized prostate cancer with prostate-specific antigen (PSA) < 0.1, or has undergone potentially curative therapy with no evidence of disease for five years, or who is deemed at low risk for recurrence by his/her treating physician.
21. Patient with central nervous system (CNS) metastases and/or carcinomatous meningitis.
22. History of gastrointestinal disease that could potentially impact the ability of the patient to swallow and/or absorb study drug (i.e., gastrointestinal surgery, malabsorption syndrome, subjects requiring the use of feeding tube)
23. History of gastrointestinal surgery or other procedures that might in the opinion of the investigator interfere with swallowing and/or absorption of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-11-19 (Actual); Primary Completion 2016-03-21 (Actual); Study Completion 2016-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise Pereria, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fenofibrate Therapy
Started | 6
Completed | 2
Not Completed | 4
Not completed — Lack of Efficacy | 4

BASELINE CHARACTERISTICS:
Arm/Group | Fenofibrate Therapy
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Rate of Response in Participants Receiving Fenofibrate Therapy
Description: To determine response rate (Strict Complete Response (sCR), Complete response (CR), Very Good Partial Response (VgPR), and Partial Response (PR)) in multiple myeloma patients receiving oral fenofibrate therapy. Response will be measured by serum and urine protein electrophoresis and immunofixation, as well as by percentage of plasma cells present on bone marrow biopsy.
Time Frame: After two cycles, about 2 months
Population: No participants achieved response to protocol therapy (Strict Complete Response (sCR), Complete response (CR), Very Good Partial Response (VgPR), or Partial Response (PR)). Two (2) patients had stable disease (SD); one (1) patient achieved Stable Disease/clinical Progressive Disease, and three (3) patients had progressive disease (PD).
Measure: Number; unit: participants
Arm/Group | Fenofibrate Therapy
Number analyzed (Participants) | 6
participants
  Strict Complete Response (sCR) | 0
  Complete response (CR) | 0
  Very Good Partial Response (VgPR) | 0
  Partial Response (PR) | 0

2. Secondary Outcome: Number of Subjects Experiencing Adverse Events
Description: To evaluate safety and tolerability of fenofibrate therapy in patients with multiple myeloma.
Time Frame: Up to 8 months
Measure: Number; unit: participants
Arm/Group | Fenofibrate Therapy
Number analyzed (Participants) | 6
participants | 5

3. Secondary Outcome: Proportion of Participants Achieving Progression-Free Survival
Description: Proportion of participants achieving progression-free survival. Measured from date of initiation of treatment (Day 1) to the earliest occurrence of any of the following events: documented disease progression, or death from any cause. Patients who are alive and progression-free will be censored at the date of last documented progression-free status.
Time Frame: 6 months, 12 months
Measure: Number; unit: participants
Arm/Group | Fenofibrate Therapy
Number analyzed (Participants) | 6
participants
  6 months | 0
  12 months | 0

ADVERSE EVENTS:
Arm/Group | Fenofibrate Therapy
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 5/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fenofibrate Therapy (N=6)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Creatinine Increased (Metabolism and nutrition disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Fatigue (General disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Flu-like Symptoms (General disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2)
Localized edema (General disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Back pain (General disorders) | 1 (1)
Bone pain (General disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Palpitations (Cardiac disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes